CLINICAL TRIAL: NCT02907398
Title: Adherence and Outcome of Upper Airway Stimulation (UAS) for OSA International Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ADHERE UAS Registry
Record Dates: First submitted 2016-08-30; First posted 2016-09-20 (Estimated); Last update posted 2025-06-19 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Neurostimulation; Hypoglossal nerve; Tongue; Upper airway stimulation; Surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ADHERE: This group will include 250 patients who have been implanted with the Inspire therapy system, enrolled in the ADHERE Registry, and are willing to complete a follow-up home sleep apnea test (HSAT).
  Interventions: Device: Inspire therapy
- CONTROL: This group will include 100 patients who have been denied insurance coverage of the Inspire therapy system implant by their provider, have had no intervention (Inspire), and are willing to complete a HSAT and provide information about their OSA treatment after denial.
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Inspire therapy
  Other Names: ADHERE
  Groups: ADHERE
Other: No intervention
  Other Names: CONTROL
  Groups: CONTROL

SUMMARY:
Inspire intends to conduct this registry to: 1) collect Inspire therapy clinical evidence in the clinical practice setting; 2) collect additional information on the effectiveness, use and safety in the commercial setting; and 3) engage physician customers to report the collective outcome within a group of properly trained programs that utilize Inspire therapy on a regular basis.

In addition, a sub-study will be conducted under this Registry at a limited number of Registry centers and will include a cohort of Registry patients and a cohort of patients who have not received the Inspire therapy device due to denial of insurance coverage. The two sub-study cohorts' quality of life and AHI data will be compared.

DETAILED DESCRIPTION:
This registry is a multi-center, prospective, observational registry, conducted in the United States and Europe. Some data may be collected retrospectively in patients currently implanted (implanted prior to enrollment) through the 12-month follow-up time frame. The CE-marked and FDA-approved Inspire system will be used within its intended use, allowing for of use of any future approved system component models. This protocol does not include any additional stressful or invasive tests, which are not a part of standard of care.

ELIGIBILITY:
Inclusion Criteria:

Any patient implanted with or receiving an Inspire implant, who meets the following criteria, is eligible to participate in the registry:

1. Capable of giving informed consent, as required per institution
2. Willing to return for routine clinic visits as required for Inspire therapy management

Exclusion Criteria:

Any patient who meets any of the following criteria will not be eligible to participate in the registry

1. Has a life expectancy of less than 1 year
2. Any reason the clinician deems patient is unfit for participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled for an Inspire implant or who had an Inspire implant prior to the initiation of the Registry. In addition, those patients who were denied insurance coverage for the implant.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Apnea Hypopnea (AHI) from Baseline to 12-Months | Baseline through 12 months
  Apnea Hypopnea Index (AHI) is a measure of OSA severity. The AHI will be determined by the AHI score at the post-titration visit compared with the pre-implant baseline score.
Change in Epworth Sleepiness Scale (ESS) from Baseline to 12 Months | Baseline through 12 months
  The Epworth Sleepiness Scale (ESS) is a validated instruction that rates a subject's daytime sleepiness. ESS scores range from 0 to 24, with a lower score indicating less daytime sleepiness. An ESS score of 10 or less is equivalent to the normalized population. The ESS efficacy endpoint will be determined by the ESS score at the 12-month follow-up as compared to baseline.

SECONDARY OUTCOMES:
Patient Experience with Therapy (PET) | Through 12 months
  The PET is a survey deigned to collect information about patients' experience with the Inspire therapy. Information will be collected once the therapy is activated about relative satisfaction with the therapy over time.
Therapy Adherence | Through 12 months
  Therapy use, reported as hours of use per week, is record by Inspire device and can be collected upon interrogation of the device in the clinic. This value can be used to quantify device use and adherence over time.
Advance or Additional Titrations | Through 12 months
  The patient will report the number of in-office or sleep lab device titrations completed.
Physical Assessment | Baseline through 12 months
  Blood pressure, and height (in either cm or in) & weight (in either kg or lbs) will be used to calculate Body Mass Index at baseline and through study completion.
Clinical Global Impression (CGI-I) | Baseline through 12 months
  The Clinical Global Impression (CGI-I) is a clinician assessment of how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. During the assessment the physician rates the patient's obstructive sleep apnea by selecting 1 of 7 categories that range from very much worse to very much improved (in comparison to baseline).
Device Data Collection | Through 12 months
  Device programming and adjustment data recorded during follow-up visits will be collected from physician and patient programmers.
Insomnia Severity Index (ISI) | Baseline through 12 months
  The Insomnia Severity Index (ISI) is a 7 item self-report instrument that measures patient perception of both nocturnal and diurnal symptoms of insomnia. Scores range from 0 to 28, with a lower score indicating less severe insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Gimmestad, Study Director — Inspire Medical Systems, Inc.
Locations (63):
- United States (52):
  - The University of Alabama for the University of Alabama at Birmingham, Birmingham, Alabama
  - Valley Sleep Center, Mesa, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Valley ENT, Scottsdale, Arizona
  - The Neurology Center of Southern California, Carlsbad, California
  - University of Southern California, Los Angeles, California
  - Stanford University Medical Center, Redwood City, California
  - University of Colorado Denver, Aurora, Colorado
  - Middlesex Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Health, Gainesville, Florida
  - Central Florida Pulmonary, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Northshore University Hospital, Glenview, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Richard L Roudebush VA Medical Center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Wayne State University, Dearborn, Michigan
  - Michigan Heart - St Joseph Mercy Health System, Ypsilanti, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Cloud Ear, Nose and Throat Clinic, Saint Cloud, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Luke's Hospital, Chesterfield, Missouri
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Long Island Jewish/Northwell Health, New Hyde Park, New York
  - Weill Cornell Medicine, New York, New York
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Sleep Management Institute, Cincinnati, Ohio
  - University Hospitals Case Western, Cleveland, Ohio
  - MetroHealth Systems, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University and Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Reading Hospital, Reading, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center/ Baptist Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Ogden Clinic, Ogden, Utah
  - Virginia Heart Center for Sleep and Wellness, Fairfax, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Puget Sound ENT, Edmonds, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- Germany (7):
  - Universitatsklinikum Hamburg Eppendorf, Hamburge, Germany
  - Technische Universitat Dresden, Dresden
  - Asklepios Klinik Harburg, Hamburg
  - University of Lubeck, Lübeck
  - Universitäts-HNO-Klinik Mannheim, Mannheim
  - Klinikum rechts der Isar der Technischen Universitat Munchen, Munich
  - Klinikum Stuttgart-Katharinenhospital, Stuttgart
- Netherlands (2):
  - OLVG, Amsterdam
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
- Kantonnspital Baselland-Liestal, Liestal, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bosschieter PFN, de Vries N, Mehra R, Manchanda S, Padhya TA, Vanderveken OM, Ravesloot MJL; ADHERE Registry Investigators. Similar effect of hypoglossal nerve stimulation for obstructive sleep apnea in 5 disease severity categories. J Clin Sleep Med. 2022 Jun 1;18(6):1657-1665. doi: 10.5664/jcsm.9956. PMID 35236551